CLINICAL TRIAL: NCT03829241
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Trial of Troriluzole in Generalized Anxiety Disorder
Brief Title: Randomized Trial of Adult Participants With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHV4157-207
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder (GAD)
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind to Sponsor, Investigator and Subject
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Troriluzole (Experimental): Randomization phase (Weeks 1 through 8): Participants received troriluzole 100 mg capsules twice daily (BID) orally for up to 8 weeks in the double-blind (DB) randomization phase.
  Extension phase (Weeks 9 through 56): Participants, who completed the randomization phase and for whom the investigator believed open-label (OL) treatment could offer an acceptable risk-benefit profile, entered the extension phase and received OL troriluzole capsules (continuing on the same dose and regimen that was taken at the end of the randomization phase) for up to additional 48 weeks.
  Interventions: Drug: Troriluzole
- Placebo (Placebo Comparator): Randomization Phase (Weeks 1 through 8): Participants received troriluzole matching placebo capsules BID orally for up to 8 weeks in the DB randomization phase.
  Extension Phase (Weeks 9 through 56): Participants, who completed the randomization phase and for whom the investigator believed OL treatment could offer an acceptable risk-benefit profile, entered the extension phase and received OL troriluzole capsules (continuing on the same dose and regimen that was taken at the end of the randomization phase) for up to additional 48 weeks.
  Interventions: Drug: Troriluzole; Drug: Placebo

INTERVENTIONS:
Drug: Troriluzole — 100 mg capsule
  Other Names: BHV-4157
Drug: Placebo — Placebo matched to troriluzole
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of troriluzole versus placebo in participants with generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of generalized anxiety disorder (GAD) either moderate or severe as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) as confirmed by the MINI at Screening, in addition to a psychiatric evaluation by a board- certified or Biohaven-approved board-eligible psychiatrist; The duration of illness must be ≥ 1 year
* Hamilton Anxiety Rating Scale (HAM-A) Total Score of ≥ 18 at both Screening and Baseline
* Clinical Global Impression of Severity Scale (CGI-S) score of ≥ 4 at both Screening and Baseline
* Determined by the investigator to be medically stable at baseline/randomization as assessed by medical history, physical examination, laboratory test results, and electrocardiogram testing. Participants must be physically able and expected to complete the trial as designed
* Minimum of 6 years of education or equivalent to complete necessary scales and understand consent forms
* Participants must be able to understand and agree to comply with the prescribed dosage regimens and procedures; report for regularly scheduled office visits; and reliably communicate with study personnel about adverse events and concomitant medications
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to dosing at Baseline

Exclusion Criteria:

* Participants with a primary DSM-V psychiatric disorder diagnosis other than GAD within the past 6-months. Note: Participants with a secondary diagnosis of comorbid social anxiety disorder or specific phobia are allowed, if in the investigator's judgement, the diagnosis is not sufficiently prominent and active so as to be confound the assessment of GAD symptoms
* Participants should be excluded at screening or baseline if any medical or psychiatric condition other than GAD, as specified in the inclusion criteria, could predominantly explain or contribute significantly to the subjects' symptoms or that could confound assessment of GAD symptoms
* Participants who report a history of inadequate response (per investigator judgement) to 3 or more adequate trials (including current trial) of any SSRI or SNRI, at an adequate dose and adequate duration (at least 8 weeks) for the treatment of GAD within the 3 years prior to randomization
* Hamilton Depression Rating Scale 17 (HAM-D-17) item 1 of >1 at Screening or Baseline
* HAM-D-17 of > 19 at Baseline
* Any eating disorder within the last 12 months prior to Screening
* Acute suicidality in the last 12 months, or suicide attempt or self-injurious behavior in the last 12 months prior to Screening
* Score of >0 on the Sheehan Suicidality Tracking Scale for the period of 12 months prior to screening, and at baseline
* History of psychosurgery, deep brain stimulation (DBS) or electroconvulsive therapy (ECT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - Woodland International Research Group, Little Rock, Arkansas
  - Axiom Research, LLC, Colton, California
  - Pharmacology Research Institute, Encino, California
  - University of California, San Francisco-Fresno, Fresno, California
  - Collaborative Neuroscience Network, LLC., Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - CalNeuro Research Group, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Research Partners, LLC, Oakland, California
  - NRC Research Institute, Orange, California
  - Desert Valley Research, Rancho Mirage, California
  - Atemis Institute for Clinical Research, San Marcos, California
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - CNS Network, Torrance, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Child Study Center at Yale University School of Medicine, New Haven, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Meridien Research, Bradenton, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Galiz Research, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - iResearch Atlanta LLC, Decatur, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Phoenix Medical Research, Prairie Village, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Boston Clinical Trials, Boston, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Altea Research Institute, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Salem, Oregon
  - Suburban Research Associates, Inc., Media, Pennsylvania
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Volunteer Research Group, an AMR Company, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Baylor College of Medicine, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 53 sites in the United States.
Pre-assignment Details: A total of 881 participants were enrolled, of which 402 participants were randomized in a 1:1: ratio to receive troriluzole or placebo. 479 participants were not randomized due to withdrawal of concent, lost to follow-up, failed inclusion/exclusion criteria, or other reasons.
Period: Randomization Phase (Week 1 to Week 8)
Arm/Group | Troriluzole | Placebo
Started | 202 | 200
Treated | 199 | 191
Modified Intent-to- Treat (mITT) Participants (Modified intent-to-treat (mITT) participants in the randomization phase included randomized participants who received at least 1 dose of blinded study drug and provided a non-missing baseline assessment and at least 1 non-missing post-baseline efficacy assessment.) | 198 | 187
Completed | 171 | 158
Not Completed | 31 | 42
Not completed — Withdrawal of Consent | 16 | 19
Not completed — Lost to Follow-up | 5 | 11
Not completed — Sponsor Request | 0 | 1
Not completed — Adverse Event | 8 | 9
Not completed — Non compliance | 2 | 1
Not completed — Pregnancy | 0 | 1
Period: Extension Phase (Week 9 up to Week 48)
Arm/Group | Troriluzole | Placebo
Started (Participants who continued into the extension phase) | 159 | 154
Treated | 153 | 149
Completed | 0 | 0
Not Completed | 159 | 154
Not completed — Withdrawal of Consent | 20 | 24
Not completed — Lost to Follow-up | 9 | 7
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Request | 117 | 108
Not completed — Significant Protocol Violation | 0 | 1
Not completed — Adverse Event | 11 | 11
Not completed — Non compliance | 1 | 1
Not completed — Pregnancy | 0 | 2

BASELINE CHARACTERISTICS:
Population: Treated participants in the randomization phase: Enrolled participants who received at least 1 dose of blinded study therapy (troriluzole or placebo).
Groups:
- Troriluzole: Randomization phase (Weeks 1 through 8): Participants received troriluzole 100 mg capsules BID orally for up to 8 weeks in the DB randomization phase.
  Extension phase (Weeks 9 through 56): Participants, who completed the randomization phase and for whom the investigator believed OL treatment could offer an acceptable risk-benefit profile, entered the extension phase and received OL troriluzole capsules (continuing on the same dose and regimen that was taken at the end of the randomization phase) for up to additional 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Troriluzole | Placebo | Total
Number analyzed (Participants) | 199 | 191 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (12.72) | 37.5 (12.59) | 38.0 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 147 | 299
  Male | 47 | 44 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 36 | 65
  Not Hispanic or Latino | 170 | 155 | 325
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 29 | 26 | 55
  White | 151 | 151 | 302
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 2 | 1 | 3
Hamilton Anxiety Rating Scale (HAM-A): Total score [Mean (Standard Deviation); unit: score on a scale] — The HAM-A is a investigator-administered scale designed to rate the severity of anxiety as well as the type of symptoms in participants with GAD. The scale consisted of 14 items: anxious mood, tension, fears, insomnia, concentration, depressed mood, behavior at interview, somatic muscular, somatic sensory, cardiovascular, respiratory, gastrointestinal, genitourinary, and autonomic symptoms. Each item was scored on a scale of 0 (not present) to 4 (severe) with a total score range of 0-56. a decreased score indicating a decrease in anxiety symptoms.
  score on a scale | 24.7 (4.34) | 24.1 (3.80) | 24.4 (4.08)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the HAM-A Total Score at Week 8
Description: The HAM-A was an investigator-administered scale and consisted of 14 items: anxious mood, tension, fears, insomnia, concentration, depressed mood, behavior at interview, somatic muscular, somatic sensory, cardiovascular, respiratory, gastrointestinal, genitourinary, and autonomic symptoms. Each item was scored on a scale of 0 (not present) to 4 (severe) with a total score range of 0-56. A decreased score indicated a decrease in anxiety symptoms.
Time Frame: Baseline, Week 8
Population: The mITT participants in the randomization phase (randomized participants who received at least 1 dose of blinded study therapy [troriluzole or placebo], and provided a non-missing baseline assessment and at least 1 non-missing post-baseline efficacy assessment during the randomization phase) were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Troriluzole: Randomization phase (Weeks 1 through 8): Participants received troriluzole 100 mg capsules BID orally for up to 8 weeks in the DB randomization phase.
- Placebo: Randomization Phase (Weeks 1 through 8): Participants received troriluzole matching placebo capsules BID orally for up to 8 weeks in the DB randomization phase.
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 198 | 187
score on a scale | -9.28 [-10.23 to -8.32] | -9.35 [-10.34 to -8.36]
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; Model-based summary statistics are from a mixed model with repeated measures, including fixed effects for treatment, visit, treatment-by-visit interaction, baseline score, baseline score-by-visit interaction as covariates, and participant as random effect; Test type: Superiority; p = 0.917, Mixed Models Analysis; LS Mean Difference = -0.07, 95% CI 2-sided [-1.45 to 1.30], Standard Error of Mean 0.70

2. Secondary Outcome: Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), TEAEs Leading to Discontinuation, and TEAEs Judged to be Related to Study Medication During Randomized Phase
Description: A serious adverse event (SAE) was defined as any event that met any of the following criteria: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received rimegepant; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention.
  Treatment-emergent AEs (TEAEs) in the randomization phase included any adverse event (AE) with an onset date on or after the first day of double-blind study drug and up to the first day of open-label study drug in the extension phase (for participants entering the extension phase) or last day of the randomization phase study drug + 30 days.
Time Frame: From first dose to Week 8 plus 30 days (maximum duration: 12 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 199 | 191
Participants
  Participants with at least 1 serious TEAE | 0 | 0
  Participants with at least 1 TEAE related to study medication | 59 | 47
  Participants with at least 1 TEAE leading to withdrawal from study drug | 11 | 11

3. Secondary Outcome: Number of Participants With Serious TEAEs, TEAEs Leading to Discontinuation, and TEAEs Judged to be Related to Study Drug During Extension Phase
Description: An SAE was defined as any event that met any of the following criteria: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received rimegepant; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention.
  TEAEs in the extension phase included any AE with an onset date on or after the first day of the study drug in the extension phase and up to the last day of the study drug in the extension phase + 30 days.
Time Frame: From Week 9 to the last dose of troriluzole in extension phase plus 30 days (maximum duration: 333 days)
Population: Treated participants in the extension phase: Treated participants in the randomization phase who received at least 1 dose of troriluzole in the open-label (OL) extension phase.
Measure: Count of Participants; unit: Participants
Groups:
- Troriluzole; Placebo: Extension phase (Weeks 9 through 56): Participants, who completed the randomization phase and for whom the investigator believed OL treatment could offer an acceptable risk-benefit profile, entered the extension phase and received OL troriluzole capsules (continuing on the same dose and regimen that was taken at the end of the randomization phase) for up to additional 48 weeks.
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 153 | 149
Participants
  Participants with at least 1 serious TEAE | 3 | 1
  Participants with at least 1 TEAE related to study medication | 29 | 27
  Participants with at least 1 TEAE leading to withdrawal from study drug | 9 | 12

4. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities During the Randomization Phase
Description: Clinically significant laboratory abnormalities were defined as Grade 3 to 4 laboratory test results according to numeric laboratory test criteria found in Common Technical Criteria for Adverse Events (CTCAE) Version 5.0 (2017) or the Division of Acquired Immune Deficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1 (2017), where Grade 3=Severe and Grade 4=Potentially Life Threatening. Laboratory test groups of clinical interest included hematology, serum chemistry, and urinalysis.
Time Frame: From first dose to Week 8 plus 30 days (maximum duration: 12 weeks)
Population: Treated participants in the randomization phase with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 194 | 178
Participants
  Hemoglobin: number analyzed (Participants) | 193 | 178
  Hemoglobin | 0 | 0
  Leukocytes: number analyzed (Participants) | 193 | 178
  Leukocytes | 0 | 0
  Lymphocytes, low: number analyzed (Participants) | 193 | 178
  Lymphocytes, low | 0 | 0
  Lymphocytes, high: number analyzed (Participants) | 193 | 178
  Lymphocytes, high | 0 | 0
  Neutrophils: number analyzed (Participants) | 193 | 178
  Neutrophils | 0 | 0
  Platelets: number analyzed (Participants) | 193 | 178
  Platelets | 0 | 0
  Alanine Aminotransferase | 1 | 0
  Albumin | 0 | 0
  Alkaline Phosphatase | 0 | 0
  Aspartate Aminotransferase | 2 | 0
  Bicarbonate | 0 | 0
  Bilirubin | 0 | 0
  Calcium, low | 0 | 0
  Calcium, high | 0 | 0
  Creatine Kinase | 3 | 1
  Creatinine | 0 | 0
  Glucose, low | 0 | 0
  Glucose, high | 1 | 0
  Lactate Dehydrogenase | 0 | 0
  Potassium, low | 0 | 0
  Potassium, high | 1 | 1
  Sodium, low | 0 | 0
  Sodium, high | 0 | 0
  Urate | 1 | 0
  Urine Glucose: number analyzed (Participants) | 194 | 177
  Urine Glucose | 0 | 0
  Urine Protein: number analyzed (Participants) | 194 | 177
  Urine Protein | 0 | 0

5. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 8
Description: The SDS was assessed in 3 domains: work/school (0-10), social life (0-10), and family life (0-10). The score from each domain was summed into a single-dimensional measure of global functional impairment (SDS total score) that ranged from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Baseline, Week 8
Population: The mITT participants in the randomization phase with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 177 | 174
score on a scale | -5.78 [-6.84 to -4.72] | -5.53 [-6.60 to -4.47]

6. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity Scale (CGI-S) Score at Week 8
Description: Participants rated on the seven-point severity of Illness with severity of wherein 1 = normal, not at all; 2= borderline ill; 3= mildly ill; 4= moderately ill; 5= markedly ill; 6= severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Week 8
Population: The mITT participants in the randomization phase were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 198 | 187
score on a scale | -1.19 [-1.35 to -1.03] | -1.21 [-1.38 to -1.04]

ADVERSE EVENTS:
Time Frame: Randmization Phase: From first dose to Week 8 plus 30 days (maximum duration: 12 weeks) Extension Phase: From Week 9 to the last dose of troriluzole in extension phase plus 30 days (maximum duration: 333 days)
Description: Randomization phase: Treated participants in the randomization phase - enrolled participants who received at least 1 dose of blinded study therapy (troriluzole or placebo).
  Extension phase: Treated participants in the extension phase - treated participants in the randomization phase who received at least 1 dose of troriluzole in the OL extension phase.
Groups:
- Troriluzole - Randomization Phase: Randomization phase (Weeks 1 through 8): Participants received troriluzole 100 mg capsules BID orally for up to 8 weeks in the DB randomization phase.
- Placebo - Randomization Phase: Randomization Phase (Weeks 1 through 8): Participants received troriluzole matching placebo capsules BID orally for up to 8 weeks in the DB randomization phase.
- Troriluzole - Randomization Phase/Troriluzole - Extension Phase: Extension phase (Weeks 9 through 56): Participants, who completed the randomization phase and for whom the investigator believed open-label (OL) treatment could offer an acceptable risk-benefit profile, entered the extension phase and received OL troriluzole capsules (continuing on the same dose and regimen that was taken at the end of the randomization phase) for up to additional 48 weeks.
- Placebo - Randomization Phase/Troriluzole - Extension Phase: Extension Phase (Weeks 9 through 56): Participants, who completed the randomization phase and for whom the investigator believed OL treatment could offer an acceptable risk-benefit profile, entered the extension phase and received OL troriluzole capsules (continuing on the same dose and regimen that was taken at the end of the randomization phase) for up to additional 48 weeks.
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase | Troriluzole - Randomization Phase/Troriluzole - Extension Phase | Placebo - Randomization Phase/Troriluzole - Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/191 | 0/153 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/191 | 3/153 | 1/149
Other Adverse Events (participants affected / at risk) | 43/199 | 36/191 | 28/153 | 30/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole - Randomization Phase (N=199) | Placebo - Randomization Phase (N=191) | Troriluzole - Randomization Phase/Troriluzole - Extension Phase (N=153) | Placebo - Randomization Phase/Troriluzole - Extension Phase (N=149)
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole - Randomization Phase (N=199) | Placebo - Randomization Phase (N=191) | Troriluzole - Randomization Phase/Troriluzole - Extension Phase (N=153) | Placebo - Randomization Phase/Troriluzole - Extension Phase (N=149)
Nausea (Gastrointestinal disorders) | 17 | 16 | 3 | 3
Headache (Nervous system disorders) | 8 | 12 | 7 | 2
Fatigue (General disorders) | 10 | 9 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 10 | 4 | 8 | 13
Nasopharyngitis (Infections and infestations) | 5 | 5 | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT03829241/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT03829241/SAP_001.pdf